CLINICAL TRIAL: NCT02564770
Title: A Retrospective Chart Review of the Use of MabThera (Rituximab) for the Treatment of Rheumatoid Arthritis (RA) in Australian Rheumatology Practice
Brief Title: A Retrospective Chart Review of MabThera (Rituximab) Treatment in Rheumatoid Arthritis (RA) Participants in Australia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Products Pty Ltd (Australia) (Unknown)
Responsible Party: Sponsor
Other Study IDs: ML28321
Record Dates: First submitted 2015-08-11; First posted 2015-10-01 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Rheumatoid arthritis (RA) participants: Participants who had been treated with rituximab for RA are reviewed retrospectively using chart review from Baseline until and their most recent visit to the rheumatologist prior to the conduct of the chart review.

SUMMARY:
This is a cross-sectional, observational study examining the factors leading to the therapeutic decision to use MabThera (rituximab) in participants with RA. Routine rheumatology clinical practice data of participants who are being or have been treated with rituximab for RA will be collected and analysed in this chart review.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to (>=) 18 years of age at the time of data collection
* RA diagnosed by a rheumatologist
* Treatment with rituximab for RA

Exclusion Criteria:

* Participants whose primary diagnosis and indication for rituximab treatment is a condition other than RA
* Participants who have been treated with an experimental agent for RA which is not currently approved for the treatment of RA in Australia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis (RA) participants who have been treated with rituximab
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Factors leading to Therapeutic decision to use rituximab | Up to end of study (approximately 1 month)

SECONDARY OUTCOMES:
Change in Erythrocyte sedimentation rate | Baseline and most recent visits (approximately 1 month)
Change in Immunoglobulin levels | Baseline and most recent visits (approximately 1 month)
Percentage of participants with positive or negative results for rheumatoid factor | Up to end of study (approximately 1 month)
Percentage of participants with positive or negative results for anti-cyclic citrullinated peptide antibody | Up to end of study (approximately 1 month)
Percentage of participants with positive or negative results for anti-nuclear antibodies | Up to end of study (approximately 1 month)
Disease activity score (DAS28) | At baseline visit (most recent visit prior to MabThera treatment) and at most recent visit prior to chart review (approximately 1 month)
Tender joint count (TJC) | At baseline visit (most recent visit prior to MabThera treatment) and at most recent visit prior to chart review (approximately 1 month)
Swollen joint count (SJC) | At baseline visit (most recent visit prior to MabThera treatment) and at most recent visit prior to chart review (approximately 1 month)
Duration of treatment with rituximab | From first dose to most recent rituximab infusion (approximately 1 month)
Change in C-reactive protein | Baseline and most recent visits (approximately 1 month)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Geelong, Victoria, Australia